CLINICAL TRIAL: NCT03635593
Title: Cannabis Oil for Chronic Non-CancEr Pain Treatment [CONCEPT] - Alpha (α): A Randomized Controlled Trial
Brief Title: Cannabis Oil for Chronic Non-Cancer Pain Treatment
Acronym: CONCEPT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Ramesh Zacharias, Medical Director, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MGD-011-20180805
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Chronic Non-cancer Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBD (Active Comparator): 10mg capsules Cannabidiol (CBD)
  Interventions: Drug: CBD
- CBD+THC (Active Comparator): 10mg capsules Cannabidiol (CBD) +THC tetrahydrocannabinol (CBD 5mg + (THC)
  Interventions: Drug: CBD+THC
- Placebo (Placebo Comparator): 10mg capsules placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CBD — Participants will be randomized to CBD 10mg capsules for 12 weeks. Participants will start with 1, CBD (10mg) capsule per day and self-titrate up to 8, 10mg CBD capsules (80mg) per day as needed.
  Arms: CBD
Drug: CBD+THC — Participants will be randomized to CBD+THC 10mg (CBD 5mg + THC) for 12 weeks. Participants will start with 1, 10mg CBD+THC (5mg+5mg) capsule per day and self- titrate up to 8, 10mg CBD+THC (5mg+5mg) capsules to a maximum of 80mg (40mg CBD + 40mg THC) per day as needed.
  Arms: CBD+THC
Other: Placebo — Participants randomized to placebo 10mg capsules for 12 weeks. Participants will start with 1, 10mg placebo capsule per day and self-titrate up to 8 10mg placebo capsules (80mg) per day.
  Arms: Placebo

SUMMARY:
Cannabis is being prescribed medically for chronic non-cancer pain despite limited evidence whether or not it works to reduce average pain in patients with chronic non-cancer pain. The cannabis plant (Cannabis sativa, Cannabis indica) consists of several hundred compounds of which, approximately 70 of which are thought to be active. The two active cannabinoids of interest in this trial are tetrahydrocannabinol (Δ9-THC) and cannabidiol (CBD). The goal of this trial is to determine whether CBD or CBD+THC reduces the average pain in participants with chronic non-cancer pain. The investigators also aim to determine whether CBD or CBD+THC is associated with a reduction in pain severity, pain interference, anxiety, depression, insomnia, opioids and use of benzodiazepines, analgesics, antidepressants, anxiolytics, or hypnotics amongst chronic non-cancer pain patients or an increase in physical functioning, physical health related role limitations, social functioning, mental functioning.

ELIGIBILITY:
Inclusion Criteria:

* Age >25
* Average pain score in past week of ≥ 4/10.

Exclusion Criteria:

* Personal history of bipolar disorder
* Personal or family history (first degree relative - parent of sibling) of psychotic disorders (e.g., schizophrenia)
* Active cancer (an individual undergoing active cancer chemotherapy, radiation or surgical treatment and is deemed to not be in remission as per an oncologist's report)
* Intention to travel internationally during the trial
* Uncontrolled diabetes (A1C > 11)
* Cannabis use in the past 4 weeks (recreational or medicinal)
* Current use of illicit drugs (e.g., cocaine)
* Current use of non-prescription opioids
* Unable to read and write in English
* Women who are currently pregnant or breast-feeding; or women of child-bearing age who plan to become pregnant during the trial period.

Min Age: 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-01-30 (Estimated)

PRIMARY OUTCOMES:
Average Pain Score | 12 weeks after Treatment (Week 16 of trial)
  Relative change in Average Pain Score measured by the Average Pain Score ( 0=No Pain and 10=Pain as bad as you can imagine) from the Numeric Rating Scale

SECONDARY OUTCOMES:
Pain Severity Score | Baseline, week 4, 8, 12 and 16
  Decrease in Pain Severity Score measured by composite of 4 pain items (worst, least, average, now with 0=No Pain and 10=Pain as bad as you can imagine) (mean severity score) from the Brief Pain Inventory
Pain Intensity Score | Baseline, week 4, 8, 12 and 16
  Improved Pain Intensity Score measured by mean of 7 severity items (general, activity, walking, work, mood, enjoyment of life, relations with others and sleep with 0=No Pain and 10=Pain as bad as you can imagine) from the Brief Pain Inventory
Physical Functioning Score | Baseline, week 4, 8, 12 and 16
  Increase in Physical Functioning Score measured by the SF-36V2. 10 items in this scale represent levels and kinds of limitations between the extremes of physical activities, including lifting and carrying groceries; climbing stairs; bending, kneeling or stooping and walking moderate distances. One self-care item is included to represent limitations in self-care activities. This scale captures both the presence and existent of physical limitations using a three-level response continuum. Low scores indicate significant limitations in performing physical activities, while high scores reflect little or no such limitations.
Mental Health Score | Baseline, week 4, 8, 12 and 16
  Increase in Mental Health (MH) Score measured by the SF-36V2. This 5-item scale includes one or more items from each of four major mental health dimensions (anxiety, depression, loss of behavioral/emotional control, and psychological wellbeing). Low scores on MH are indicative of frequent feelings of nervousness and depression, while high scores indicate feelings of peace, happiness, and calm all or most of the time.
Social Functioning Score | Baseline, week 4, 8, 12 and 16
  Increase in Social Functioning (SF) Score measured by the SF-36V2. This 2-item scale assesses health-related effects on quantity and quality of social activities, asking specifically either physical or emotional problems on social activities. The degree to which physical and emotional problems interfere with normal social actives increases with decreasing SF scores. The lowest score is related to extreme or frequent interference with normal social actives due to physical and emotional problems; the highest score indicates that the individual performs normal social activities without interference from physical or emotional problems..
Physical Health-related Role Limitations | Baseline, week 4, 8, 12 and 16
  Decrease in Physical Health-related Role Limitations measured by the SF-36V2. This 4-item scale covers an array of physical health-related role limitations, including a) limitations in the kind of work or other usual activities, b) reduction in the amount of time spend on work or other usual activities, c) difficulty performing work or other usual activities, and d) accomplishing less. Low scores on this scale reflect problems with work or other actives as a result of physical problems. High scores indicate little or no problems with work or other daily activities.
Depression Score | Baseline, week 4, 8, 12 and 16
  Improvement in Depression score measured by the Patient Health Questionnaire (PHQ-9). The PHQ-9 depression severity is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively. PHQ-9 total score for the nine items ranges from 0 to 27. Scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively.
Anxiety Score | Baseline, week 4, 8, 12 and 16
  Improvement in Depression score measured by the Generalized Anxiety Disorder (GAD-7). This is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively. GAD-7 total score for the seven items ranges from 0 to 21. Scores of 5, 10, and 15 represent cutpoints for mild, moderate, and severe anxiety, respectively.
Sleep Quality | Baseline, week 4, 8, 12 and 16
  Improvement in the Sleep Quality Score measured by the Insomnia Severity Index (ISI).Improvement in the Sleep Quality Score measured by the Insomnia Severity Index (ISI). Seven question added to get total score (0-28). Score of 0-7 has no clinically significant insomnia, 8-14 subthreshold insomnia, 15-21 clinical insomnia - moderate severity and 22-28 clinical insomnia - severe.
Pain Medication | Baseline, week 4, 8, 12 and 16
  Decrease in prescription pain medication use. Measured by recording initial and changes in prescription medication names, dose and frequency
Other non-pain prescription medications | Baseline, week 4, 8, 12 and 16
  Decrease in other no-pain prescription medications. Measured by recording initial and changes in non-prescription medications names, dose and frequency
Average Pain Score | Baseline, week 4, 8 and 12
  Relative change in Average Pain Score measured by the Average Pain Score ( 0=No Pain and 10=Pain as bad as you can imagine) from the Numeric Rating Scale

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Michael G. DeGroote Pain Clinic, Hamilton, Ontario
  - Toronto Poly Clinic, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No